CLINICAL TRIAL: NCT05311852
Title: Effects of Palmitoylethanolamide Co-ultramicronized With Luteoline (Pea-lut) on Frontal Lobe Functions and GABAergic Transmission in Long Covid Patients. An 8-week Randomized Controlled Trial.
Brief Title: Effects of PEA-LUT on Frontal Lobe Functions and GABAergic Transmission in Long-Covid Patients
Acronym: PL-PC19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Neurorehabilitation, Hospital of Vipiteno-Sterzing (BZ) Italy (Network)
Collaborators: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Paola Ortelli, PsyD, Principal Investigator, Department of Neurorehabilitation, Hospital of Vipiteno-Sterzing (BZ) Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEA-LUT-in-Post-Covid-19
Record Dates: First submitted 2022-03-30; First posted 2022-04-05 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Fatigue; Cognitive Deficit; COVID-19; Neurophysiologic Abnormality
Keywords: fatigue; cognitive deficits; post-covid19 syndrome
MeSH Terms: conditions — Fatigue; Cognition Disorders; COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomized and assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Masking Description: This is a double-blind randomized placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEA-LUT (Experimental): patients were required to assume granulated PEA-LUT 700/70 mg, 2 time/day for 8 weeks
  Interventions: Dietary Supplement: palmitoylethanolamide co-ultramicronized with antioxidant flavonoid luteolin (PEA-LUT)
- Placebo (Placebo Comparator): patients were required to assume granulated placebo, 2 time/day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: palmitoylethanolamide co-ultramicronized with antioxidant flavonoid luteolin (PEA-LUT) — assumption of the product at dosage of 700/70 mg 2 time/day for 8 weeks
  Arms: PEA-LUT
Dietary Supplement: Placebo — assumption of a placebo product 2 time/day for 8 weeks
  Arms: Placebo

SUMMARY:
The study explore the efficacy of PEA-LUT in patients suffering from neurological symptoms of Long-Covid

DETAILED DESCRIPTION:
Aim of this study was testing the possible therapeutic effects of an 8-week therapy with PEA-LUT on GABAB-ergic neurotransmission, LTP-like synaptic plasticity, indexed with transient potentiation of motor evoked potentials (MEP) amplitude after repetitive TMS given as intermittent theta burst stimulation (iTBS) in long COVID patients with cognitive complaints and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of SARS-CoV-2 infection confirmed through detection of virus RNA by polymerase chain reaction (PCR) testing of a nasopharyngeal swab;
* subsequent recovery from infection as defined by two consecutive negative PCR tests separated by at least a day;
* mild form of COVID-19 (symptoms may include fever, cough, sore throat, malaise, myalgia, anorexia, nausea, diarrhoea, anosmia and ageusia) without necessitating hospital admission;
* complaints of cognitive difficulties and/or sense of fatigue, persisting after SARS-CoV-2 infection.

Exclusion Criteria:

* prior or concurrent diagnosis of neurological, psychiatric, endocrine, metabolic or cardiopulmonary conditions;
* clinical and/or radiological evidence of COVID-19 related pneumonia during the active phase of the disease;
* anaemia;
* current pharmacological treatment with corticosteroids, antihistamines, antihypertensives, diuretics, antidepressants, anxiolytic or hypnotic drugs at the time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
changes in % of test amplitude in LICI 100 | LICI 100 was assessed two times, at enrollment and after 8 weeks of treatment duration
  changes % of test amplitude in long-interval intracortical inhibition, indexing intracortical GABAB-ergic, transmission, are expected

SECONDARY OUTCOMES:
changes in % of test amplitude in SAI 20 | SAI 20 was assessed two times, at enrollment and after 8 weeks of treatment duration
  changes % of test amplitude in short-latency afferent inhibition, to evaluate M1 inhibition induced by sensory afferents, are expected
change in LTP-like cortical plasticity | LTP-like cortical plasticity was assessed at two times, at enrollment and after 8 weeks of treatment duration
  change of MEP modulation after intermittent theta burst stimulation (iTBS)

OTHER OUTCOMES:
changes in Montreal Cognitive Assessment score | Montreal Cognitive Assessment was assessed at enrollment and after 8 weeks of treatment duration
  changes in Montreal Cognitive Assessment score, for evaluating the global cognition, are expected
changes in Frontal Assessment Battery score | Frontal Assessment Battery was assessed at enrollment and after 8 weeks of treatment duration
  changes in Frontal Assessment Battery score, for evaluating the executive functions, are expected

CONTACTS AND LOCATIONS:
Overall Officials: Leopold Saltuari, Md, Study Director — Department of Neurorehabiliation - Hospital of Vipiteno-Sterzing
Locations (1):
- Hospital of Vipiteno-Sterzing, Sterzing, BZ, Italy